CLINICAL TRIAL: NCT05438615
Title: A Prospective Study to Compare Lenses Having Two Different Proximity Control Designs for Overnight Wear for Treatment of Naturally Occurring Myopia From -4 to -6 Diopters Sphere With Refractive Astigmatism up to -1.75 Diopters
Brief Title: Corneal Refractive Therapy Design Comparison for -4 to -6 Diopter Treatment for Overnight Wear for Myopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015W0189
Record Dates: First submitted 2015-12-17; First posted 2022-06-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2022-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corneal Refractive Therapy - spherical (Experimental): Subjects eyes shall be treated with two pair of the proximity control lenses in Paragon paflufocon D material by the qualified clinical investigator. The subjects shall be randomized for which of the two designs are applied first. The first pair shall be dispensed and follow-up examinations shall be conducted at 1 day, 1 week, and 2 weeks. Each subject shall then cease wearing lenses for at least 7 days and be re-examined to determine that the corneal curvature has returned to its baseline measure. The second design shall be dispensed and follow-up examinations shall be conducted at 1 day, 1 week, and 2 weeks. Each subject shall then cease wearing lenses for at least 7 days and be re-examined to determine that the corneal curvature has returned to its baseline measure.
  Interventions: Other: Corneal Refractive Therapy-spherical
- Corneal Refractive Therapy - aspherical (Experimental): Subjects eyes shall be treated with two pair of the proximity control lenses in Paragon paflufocon D material by the qualified clinical investigator. The subjects shall be randomized for which of the two designs are applied first. The first pair shall be dispensed and follow-up examinations shall be conducted at 1 day, 1 week, and 2 weeks. Each subject shall then cease wearing lenses for at least 7 days and be re-examined to determine that the corneal curvature has returned to its baseline measure. The second design shall be dispensed and follow-up examinations shall be conducted at 1 day, 1 week, and 2 weeks. Each subject shall then cease wearing lenses for at least 7 days and be re-examined to determine that the corneal curvature has returned to its baseline measure.
  Interventions: Other: Corneal Refractive Therapy-aspherical

INTERVENTIONS:
Other: Corneal Refractive Therapy-spherical — A comparison of two different designs of Corneal Refractive Therapy contact lenses will be done. Each will be worn for two weeks. The sponsor will mask which lens will be first or second in the trial.
  Arms: Corneal Refractive Therapy - spherical
Other: Corneal Refractive Therapy-aspherical — A comparison of two different designs of Corneal Refractive Therapy contact lenses will be done. Each will be worn for two weeks. The sponsor will mask which lens will be first or second in the trial.
  Arms: Corneal Refractive Therapy - aspherical

SUMMARY:
The primary objective of this study is to compare the effectiveness of two proximity control geometry lens designs to treat eyes with pretreatment myopia between -4.00 and -6.00 D myopia with and without refractive astigmatism in a modality involving overnight wearing.

DETAILED DESCRIPTION:
Each subject shall undergo a comprehensive eye examination to determine eligibility. Subjects must meet all eligibility criteria. All eyes shall be treated with two pair of the proximity control lenses by the qualified clinical investigator. The first pair shall be dispensed and scheduled follow-up examinations shall be conducted at one day, one week, and two weeks after dispensing lenses. Each subject shall then cease wearing lenses for at least 7 days and be re-examined to determine that the corneal curvature has returned to its baseline measure. The second design shall be dispensed and scheduled follow-up examinations shall be conducted at one day, one week, and two weeks after dispensing lenses. Each subject shall then cease wearing lenses for at least 7 days and be re-examined to determine that the corneal curvature has returned to its baseline measure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients may be male or female, of any race, and at least 18 years old at the time of the pre-treatment examination.
2. The prospective eye(s) must have naturally occurring refractive myopia from -4.00 to -6.00 diopters sphere (spectacle plane), with up to -1.75 diopters of refractive astigmatism (spectacle plane), as determined by manifest refraction (phoropter or trial frame with a 12.5 mm vertex distance).
3. Patients must have best spectacle corrected visual acuity of at least 0.04 logMAR in each eye.
4. If the Subject wears rigid contact lenses in the prospective eye(s), lens use must cease at least four (4) weeks prior to the pre-treatment examination. The subject must have two central keratometry readings taken that are at least one week apart. The two readings shall not differ by more than 0.50 diopter in either meridian. The mires should be regular.
5. Patients must be willing and capable to return for all scheduled follow-up visits for a period of at least 6 months.

Exclusion Criteria:

1. Female patients who are pregnant, breast-feeding or intend to become pregnant over the course of the study.
2. Patients with a history of any of the following medical conditions: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to active thyroid disorders and diabetes), lupus, and rheumatoid arthritis.

   Note: The presence of diabetes (either type 1 or 2), regardless of disease duration, severity or control, shall specifically exclude patients from eligibility.
3. Patients with a history of intraocular or corneal surgery (including cataract extraction), active ophthalmic disease or abnormality (including, but not limited to, blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization >1mm from limbus), clinically significant lens opacity, clinical evidence of trauma (including scarring).

   Note: This includes any Subject with open angle glaucoma, regardless of medication regimen or control. Additionally, any Subject with an intraocular greater than 21 mm Hg at baseline is specifically excluded from eligibility.
4. Patients with evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye.
5. Patients with pupil size greater than 5.5 mm in photopic illumination as measured with infrared pupillometry, pupil detection component of computer assisted video keratography, or slit lamp reticule.
6. Patients who are participating in any other clinical trial (FDA or other).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10-27 (Actual); Study Completion 2016-10-27 (Actual)

PRIMARY OUTCOMES:
Refraction | Two weeks after successful fitting of each lens
visual acuity | Two weeks after successful fitting of each lens

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Barr, OD MS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States